CLINICAL TRIAL: NCT05538715
Title: Comperative Clinical, Microcircular, Surface Scanning, Radiological and Histological Evaluation of Two Different Flap Techniques - A Prospective Randomized Clinical Trial/
Brief Title: Reconstruction of Localized Alveolar Ridge Defects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Collaborators: Geistlich Pharma AG (Industry); Institut Straumann AG (Industry); Dicomlab Kft. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Augmentation-Semmelweis-Perio
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-09

CONDITIONS: Partial-edentulism
Keywords: guided surgery; xenogenic graft; augmentation; surface scanning; Laser Speckle Contrast Imaging

STUDY DESIGN:
Intervention Model Description: Test group: Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a full-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
  Control group: Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a split-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not aware of the randomly assigned flap design. Independent examiners are not aware of patient allocation during analysis of clinical and radiographic data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Split-thickness group (Experimental): Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a split-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
  Interventions: Procedure: Split-thickness group
- Full-thickness group (Experimental): Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a full-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
  Interventions: Procedure: Full-thickness group

INTERVENTIONS:
Procedure: Split-thickness group — Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a split-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
  Arms: Split-thickness group
Procedure: Full-thickness group — Following randomization, horizontal guided bone regeneration utilizing Bio-Oss (Geistlich, Wolhusen, Switzerland) and autogenous bone in combination with Bio-Gide membrane (Geistlich, Wolhusen, Switzerland). Surgery is performed with a full-thickness flap design in the posterior maxilla or mandible in partially edentolous patients.
  Arms: Full-thickness group

SUMMARY:
The aim of the present prospective randomized controlled study is to compare the clinical, radiological, micro-circulation, and histology of a novel, semi-thick, and conventional full-thickness mucoperiosteal flap technique during horizontal alveolar ridge augmentation.

DETAILED DESCRIPTION:
The aim of our study was to compare the clinical, radiological, circulatory, and histological studies of a novel, split-thickness and conventional full-thickness mucoperiosteal flap technique during horizontal alveolar ridge augmentation surgeries. Flap formation was performed in the test group using the novel split-thickness surgical technique, and in the control group using the full-thickness mucoperostatial surgical technique. The novel split-thickness flap technique to be studied results in a predictable, closed healing based on our preliminary results, thus ensuring the conditions for successful augmentation. We primarily want to investigate what hard and soft tissue changes result from ridge augmentation with a novel split-thickness flap technique after 6 months, compared to a surgical technique based on full thick flap formation accepted as a standard procedure in the literature. Our secondary examination methods: examination of early wound healing and micro-circulation after augmentation interventions by LSCI method; histological evaluation at prosthetically designed implant positions.

ELIGIBILITY:
Inclusion Criteria:

* at least one edentulous maxillary/mandibulary premolar or molar site with horizontal bone loss
* full- mouth plaque and bleeding scores (FMPS and FMBS) <20%
* good patient compliance (including willingness to participate in the follow-up procedures) signed informed consent-

Exclusion Criteria:

* Active infectious diseases (HBV, HCV, HIV, TB, SARS CoV-2, etc.)
* Current chemotherapy or radiotherapy
* Radiation treatment of the former head and neck region (not older than 2 years)
* Untreated insulin-dependent diabetes mellitus
* Clinically significant osteoporosis or other systemic disease affecting bone metabolism
* Clinically significant circulatory disorders such as decompensated cardiac failure
* Haemodynamically significant heart failure or myocardial infarction within the last 3 months
* Clinically significant coagulation disorder
* Current or previous systemic corticosteroid therapy (not older than 2 months)
* Current or previous systemic bisphosphonate therapy
* Pregnant or breastfeeding mothers
* Smoking
* Drug addiction, alcoholism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Orovestibular ridge width | 6 months postoperatively
  On prealigned pre- and postoperative CBCT cross-sections, linear measurements were taken parallel to a reference base to determine the orovestibular width of the surgical area.
Dimensional change of keratinized Gingiva | 6 months postoperatively
  Pre-and postoperatively a surface scan is performed using a Planmeca Emerald intraroral scanner. The superimposition of the measurements was used to evaluate the soft tissue changes associated with the treatments in 3 dimension.

SECONDARY OUTCOMES:
Histomorphometrical analysis | Following reentry 6 months after augmentation
  Percentage of newly formed bone, bone substitute and connective tissue
Gingival blood flow measurement at the early wound healing phase | Pre-operative and 1, 3, 5, 7, 10, 14, 21, 28 days and 2, 3, 4, 5 and 6 months after surgeries.
  Investigation of pre- and postoperative gingival blood flow using Laser Speckle Contrast Imager.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Somodi K, Dobos A, Bartha F, Solyom E, Windisch P, Palkovics D, Molnar B. Changes in soft tissue dimensions following horizontal guided bone regeneration with a split-thickness flap design - evaluation of 8 cases with a digital method. Head Face Med. 2024 Sep 28;20(1):53. doi: 10.1186/s13005-024-00456-8. PMID 39342334